CLINICAL TRIAL: NCT01611649
Title: Profilo Degli Acidi Grassi Omega-3 Dei Globuli Rossi in Neonati Sani Alimentati Con Una Formula Per l'Infanzia Contenente Una Miscela di Grassi Del Latte e Oli Vegetali
Brief Title: Effect of a Mix of Dairy Lipids and Plant Oils in Infant Formula on Omega-3 Fatty Acid in Red Blood Cells
Acronym: REBECA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lactalis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LRD-2012-REBECA
Record Dates: First submitted 2012-05-25; First posted 2012-06-05 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Infant Development
Keywords: infant formula; dairy lipids; omega-3
MeSH Terms: interventions — Plant Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dairy lipids and plant oils (Experimental)
  Interventions: Dietary Supplement: Formula containing dairy lipids and plant oils
- Plant oils (Experimental)
  Interventions: Dietary Supplement: Formula containing plant oils
- Dairy lipids and plant oils, DHA+ARA (Experimental): DHA: docosahexaenoic acid, ARA: arachidonic acid
  Interventions: Dietary Supplement: Formula containing dairy lipids and plant oils, DHA+ARA
- Human milk (No Intervention)

INTERVENTIONS:
Dietary Supplement: Formula containing dairy lipids and plant oils — 4 months consumption
  Arms: Dairy lipids and plant oils
Dietary Supplement: Formula containing plant oils — 4 months consumption
  Arms: Plant oils
Dietary Supplement: Formula containing dairy lipids and plant oils, DHA+ARA — 4 months consumption, DHA+ARA supplemented formula containing dairy lipids and plant oils
  Arms: Dairy lipids and plant oils, DHA+ARA

SUMMARY:
The objective of this study is to determine whether the use of a mix of dairy lipids and plant oils in infant formula can increase the sum of omega-3 fatty acids levels in membrane phospholipids of red blood cells (RBC) in 4 month-old infants compared with a formula containing only lipids of plant origin.

ELIGIBILITY:
Inclusion Criteria:

* Full term healthy newborn from normal pregnancy
* Newborn whose mother decided to not breastfeed or to stop breastfeed before the third week of life

Exclusion Criteria:

* Newborn with low-birth-weight (<2500 g)
* Newborn whose parents have planned a move within 6 months after birth
* Family history of allergy to milk protein

Max Age: 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Sum of omega-3 fatty acid levels in membrane phospholipids of RBC | after 4 months of consumption
  alpha linolenic acid (ALA) + eicosapentaenoic acid (EPA) + docosapentaenoic acid (DPA) + docosahexaenoic acid (DHA)

SECONDARY OUTCOMES:
Serum total fatty acid levels | after 4 months of consumption
Insulin-like Growth Factor 1 (IGF1) blood levels | after 4 months of consumption
Lipid profile (triglyceride, high-density lipoprotein HDL, low-density lipoprotein LDL, total cholesterol) | after 4 months of consumption
Amount of formula consumed, occurrence of spit-up and vomit, description of the number, color and consistency of infant stools as a measure of tolerance to the formula | during the 4 months consumption period
Growth parameters: weight, height, head circumference and body composition: amount of lean and fat mass | during the 4 months consumption period
Total fatty acid levels in membrane phospholipids of RBC | after 4 months of consumption
Evolution of blood total fatty acids levels between 0 and 4 months | between 0 and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Mosca, Prof., Principal Investigator — Fondazione IRCCS Cà Grande Ospedale Maggiore Policlinico; Pascale le Ruyet, Dr., Study Director — Lactalis
Locations (1):
- Clinica Mangiagalli, Milan, Italy

REFERENCES:
- [Derived] Gianni ML, Roggero P, Baudry C, Fressange-Mazda C, Galli C, Agostoni C, le Ruyet P, Mosca F. An infant formula containing dairy lipids increased red blood cell membrane Omega 3 fatty acids in 4 month-old healthy newborns: a randomized controlled trial. BMC Pediatr. 2018 Feb 13;18(1):53. doi: 10.1186/s12887-018-1047-5. PMID 29433457
- [Derived] Gianni ML, Roggero P, Baudry C, Fressange-Mazda C, le Ruyet P, Mosca F. No effect of adding dairy lipids or long chain polyunsaturated fatty acids on formula tolerance and growth in full term infants: a randomized controlled trial. BMC Pediatr. 2018 Jan 22;18(1):10. doi: 10.1186/s12887-018-0985-2. PMID 29357820
- [Derived] Gianni ML, Roggero P, Baudry C, Ligneul A, Morniroli D, Garbarino F, le Ruyet P, Mosca F. The influence of a formula supplemented with dairy lipids and plant oils on the erythrocyte membrane omega-3 fatty acid profile in healthy full-term infants: a double-blind randomized controlled trial. BMC Pediatr. 2012 Oct 17;12:164. doi: 10.1186/1471-2431-12-164. PMID 23072617